CLINICAL TRIAL: NCT03385122
Title: Environmental Pollution and Health of Corinth Region. Corinthia Study
Brief Title: Environment and Cardiovascular Disease: The Corinthia Study
Status: Recruiting | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Dimitris Tousoulis, Professor of Cardiology, National and Kapodistrian University of Athens
Other Study IDs: Corinthia
Record Dates: First submitted 2017-11-20; First posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Environmental factors constitute an important but underappreciated risk factor towards the development and progression of cardiovascular disease (CVD). Environmental exposure in variable pollutants is implicated in the derangement or propagation of adverse pathophysiological processes linked with atherosclerosis, including genetic, hemodynamic, metabolic, oxidative and inflammation parameters. However no data exists concerning environmental pollution in rural or semi-rural areas. Therefore the purpose of the "Corinthia" study is to examine the impact of environmental pollution in indices of cardiovascular morbidity and mortality in a cross-sectional and longitudinal design. Corinthia study began in October 2015 and is planned to recruit 2400 individuals from different regions of Corinthia country with different environmental exposure to pollutants and different patterns of soil-ground and/or air pollution until September 2018. Baseline measurements will include lifestyle measurements, anthropometric characteristics and a comprehensive cardiovascular examination. The follow-up is planned to extent, prospectively, up to 10 years and this study is anticipated to provide valuable data on the distinct impact of soil and air pollution in early markers of atherosclerosis and cardiovascular disease and in the overall impact of environment pollution to cardiovascular morbidity and mortality.

DETAILED DESCRIPTION:
Introduction

Despite major advances in cardiovascular (CV) medicine during the last decades, deaths and morbidity from cardiovascular diseases (CVD) are increasing globally [1, 2]. It seems that population aging and population growth balances out the decline in age-specific death rates from CVD that could be attributed to more effective prevention and treatment strategies [2].

Interestingly, the progress in confronting CVD is evident around the world but notably heterogeneous. Regions with the fastest growing population dynamics experienced relative increase in CV deaths in line with global trends. In contrast, developed regions reported no detectable change or little decrease in CV mortality as rapid aging of the population offsets the declines in age-specific death rates [3]. Residual CV risk beyond traditional risk factors should be reassessed and further explored in the quest of new underlying mechanisms that could provide the substrate for innovative preventive interventions and therapeutic goals.

Under this prism, environmental factors constitute an important but underappreciated risk factor towards the development and progression of CVD [4]. Environmental exposure in variable pollutants is implicated in the derangement or propagation of adverse pathophysiological processes linked with atherosclerosis, including genetic, hemodynamic, metabolic, oxidative and inflammation parameters [4]. Recent studies suggest that chronic environmental stress is an important determinant of CVD risk, even below current regulatory standards for exposure levels [4, 5].

One of the most important studies in the field of environmental cardiology, the Multi-Ethnic Study of Atherosclerosis and Air Pollution (MESA Air) investigated the association between long-term air pollution exposure and the progression of subclinical atherosclerosis and the incidence of CVD at an urban dwelling population [6]. However no data exists concerning environmental pollution in rural or semi-rural areas. Therefore the purpose of the "Corinthia" study is to examine the impact of environmental pollution in indices of CV morbidity and mortality in a cross-sectional and longitudinal design.

Rational of the study National-based data for Greece concerning environment pollution and CVD morbidity and mortality are markedly scarce. Research activity has focused on soil and groundwater anthropogenic contamination in river basin of heavy polluted industrialized areas but without reporting associations with CVD [7]. Moreover, certain prospective or retrospective studies have examined the association of long-term exposure to air pollution with CVD morbidity in urban population [8, 9]. The region of Corinth has rural or semi-rural areas with high exposure to soil and air contamination in distinct territories-patterns. The investigators hypothesized that long term exposure to environmental pollutants mediates detrimental epigenetic, oxidative, inflammatory and pro-atherogenic effects that could accelerate the progress and the severity of CVD as well as the quality of life and the overall morbidity and mortality. Therefore, the investigators sought to investigate in a cross sectional and longitudinal design the impact of different type of environmental pollution in indices of subclinical atherosclerosis, on rates of CV morbidity and mortality and on CVD risk.

Hypothesis of the study I. The primary hypothesis of the study is that individual exposed to different environmental pollutants have increased rate of all-cause mortality.

II. The secondary hypothesis of the study is that individuals exposed to different environmental pollutants have increased rate of CV mortality and increased incidence of non-fatal CVD (i.e. acute coronary syndromes, peripheral aortic disease, cerebrovascular disease).

III. Additional hypothesis of the study is that:

1. Individuals exposed to different environmental pollutants present an adverse cardiometabolic profile in terms of surrogate markers of early atherosclerosis and oxidative stress
2. Environmental pollution affects adversely the quality of life in exposed subjects
3. Environmental pollution confers epigenetic alterations (telomere shortening, microRNAs mobilization and circulation) in subjects exposed to different pollutants

Experimental details and design of the Corinthia study The present study began at October 2015 and is planned to recruit 1500 individuals from different regions of Corinth with different environmental exposure to pollutants and different patterns of soil-ground and/or air pollution until December 2016.

The investigators plan to recruit individuals living in three different areas according to environmental pollution (Figure 1):

i. Subjects living in areas with no evidence of soil/ground or air pollution ii. Subjects living in areas with air pollution iii. Subjects living in areas with soil/ground pollution Residents of the selected regions who are not planning to move within the next 10 years will be approached. An acceptance rate of participation of approximately 80% of those eligible subjects is anticipated. Exclusion criteria for the study would be

1. Inability and unwillingness to obtain informed consent
2. Individuals less than 40 years of age The recruitment into Corinthia study will be community-based, with an emphasis on balancing recruitment across the three areas, census blocks, age categories (per decades) and gender. The sampling frame will implement information from the latest national Census and will proceed along geographic boundaries. As sampling unit we will use each household, with a goal of including no more than 2 eligible participants from different households per census block. Initial contact will be performed by telephone or door-to-door. Telephone recruitment will be based on a list built from the specified geographic boundaries. Initial contact included a screening questionnaire and household enumeration of all eligible persons. The recruitment goal is 500 participants from each of the three areas of interest. During this period the research team will communicate with the local authorities and with health services in the areas of research in order to organize the volunteering selection of the participants in each area. Responsibility of the research team is also the organization of the places where field research will take place. Pilot measurements will take place and accordingly the research team will estimate the validity of the tests, and will calculate variability coefficients of the tests.

The first 24 months will be devoted to recruitment (October 2015- September 2018).

Quality Control and repeatability of measures The research fellow recruited for the study will perform all vascular and anthropometric measurements. The research fellow will undergo a 2 month training and accreditation for these measurements. Echocardiographic measurements will be performed by the same trained cardiac physiologist.

Study Measurements Baseline measurements for participants in the "Corinthia" Study will include parameters affecting the everyday lifestyle such as smoking habits, physical activity and diet. Anthropometric (height, weight, waist circumference) socio-economic and lifestyle characteristics (marital status, educational level, economic and professional status), as well as, family history and history of cardiovascular risk factors and diseases will be recorded. The investigators also planning to identify the psychological state of individuals (using a valid Depression Scale ZUNG) and participants mental status (MMSE-Mini Mental State Examination). We will record the presence and the treatment in use, if any, of hypertension, diabetes mellitus and hypercholesterolemia. Subjects will be submitted to a full cardiac examination, including physical examination, electrocardiography, echocardiography (Evaluation of left ventricle ejection fraction, of left ventricle dimensions, evaluation of valvular function, of transmittal flow pattern, of right ventricle systolic pressure, of aortic distensibility etc.), blood pressure measurements, arterial wall properties measurement with non-invasive estimation of pulse wave velocity and estimation of atherosclerotic burden with evaluation of carotid intima media thickens and of atherosclerotic plaques in carotid arteries. Peripheral blood samples will be gathered for DNA analysis, routine biochemical tests and measurement of inflammatory markers and markers of oxidative stress. Subsequent examinations, which will include repetitions of certain baseline measurements as well as new measures, will be scheduled at approximately adjacent 2-year intervals.

Selection of regions-Environmental measurements Data on soil/ground contamination with pollutants (pesticides, fertilizers etc) and of air pollution from industrial gasses and exposures will be provided from records and measurements of the Faculty of Geology and Geoenvironment and the faculty of Environmental Physics of the National and Kapodistrian University of Athens.

Follow-up The study investigators will prospectively perform the 5 and 10-year follow-up about participants': (a) Vital status (death from any cause or due to CVD), (b) development of coronary heart disease (CHD) (i.e., myocardial infarction, angina pectoris, other identified forms of ischemia, heart failure of different types, and chronic arrhythmias) and (c) development of cerebrovascular disease.

With an anticipated loss to follow-up of approximately~15% [10] the ten year follow up data are expected to decipher the effect of long term exposure to pollution on overall and cardiovascular mortality and morbidity as well as on interim endpoints of surrogate markers of subclinical atherosclerosis. Respectively, with a type I error predefined to 0.05 and all considered to be 2-tailed, a sample size of 1500 subjects would yield adequate power (>80%) to detect a 1.5- fold change in Hazzard ratio per area-group change in the aforementioned index variable towards the secondary endpoint (all-cause mortality) taking into account an event rate of 6%, a follow up period of minimum 60 months and an anticipated loss to follow up of less than 15%. Type I error was predefined at 0.05 and all tests were considered to be 2-tailed.

Conclusion The Corinthia study is an epidemiological study of Environmental importance with a cross-sectional and prospective longitudinal design planning to provide data on the distinct impact of soil and air pollution in indices of cardiovascular morbidity and mortality and in the overall health status of a rural or semi-rural population of the Greek country.

ELIGIBILITY:
Inclusion Criteria:

* Inhabitants of Corinthia Region

Exclusion Criteria:

* Inability and unwillingness to obtain informed consent
* Individuals less than 40 years of age

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to recruit individuals living in three different areas according to environmental pollution i. Subjects living in areas with no evidence of soil/ground or air pollution ii. Subjects living in areas with air pollution iii. Subjects living in areas with soil/ground pollution
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2015-10-20 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 15 Years
  Cardiovascular death, non fatal acute myocardial infarction, non fatal stroke

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Tousoulis, Study Chair — National and Kapodistrian University of Athens, Greece, First Cardiology Clinic, Hippokratio Hospital
Locations (2):
- Greece (2):
  - 1st Cardiology Department, Hippokration General Hospital, Athens, Attica
  - Hippokration Hospital, First Cardiology Clinic, Athens

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oikonomou E, Lazaros G, Georgiopoulos G, Christoforatou E, Papamikroulis GA, Vogiatzi G, Chasikidis C, Zacharia E, Giannaki A, Bourouki E, Mavratzas T, Stofa E, Papakonstantinou M, Tousouli M, Tousoulis D. Environment and cardiovascular disease: rationale of the Corinthia study. Hellenic J Cardiol. 2016 May-Jun;57(3):194-197. doi: 10.1016/j.hjc.2016.06.001. Epub 2016 Jun 23. PMID 27451913